CLINICAL TRIAL: NCT04713917
Title: Prospective Evaluation of Innovative Therapeutic Approaches of Vaginal and Sexual Dysfunction After Breast Cancer Treatment : a Randomized Multicenter Controlled Trial
Brief Title: Evaluation of Innovative Therapeutic Approaches of Vaginal and Sexual Dysfunction After Breast Cancer Treatment
Acronym: EPIONE-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INTERmedic (Unknown); Laboratoires Vivacy (Industry); Laboratoires IPRAD PHARMA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P170927J; 2018-A01678-47 (Other: N° IDRCB)
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Locoregional and systemic treatment; Vulvovaginal atrophy; Sexual quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Lasers, Gas

STUDY DESIGN:
Intervention Model Description: An open-label multicentre controlled trial randomized in 3 parallel groups (1:1:1) :
  * Bio physical inductor : CO2 laser
  * Standard treatment : Hyaluronic Acid gel
  * Chemical bio inductor : injection of Hyaluronic Acid
Who Masked: Outcomes Assessor
Masking Description: According to the center's organization, an operator and an investigator-evaluator will be identified for each patient or for all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gel Group (Active Comparator): Two applications of HA gel (Mucogyne®) per week during one year.
  Interventions: Device: Hyaluronique Acid Gel
- Laser Group (Experimental): Laser CO2 for vulvovaginal area during 2 sessions (15 min) at visits D0 and M6.
  Interventions: Device: Laser CO2
- HA Injection Group (Experimental): Injection of 1 mL of HA at D0 and M6 (DESIRIAL®).
  Interventions: Device: Hyaluronique Acid Injection

INTERVENTIONS:
Device: Hyaluronique Acid Gel — Vaginal gel based on HA with liposomal structure applicated 2 times a week
  Arms: Gel Group
Device: Laser CO2 — The laser energy delivered along the vaginal wall heats the tissue without damaging it.
  Arms: Laser Group
Device: Hyaluronique Acid Injection — HA injection performed under the mucosae (2-3mm in depth) following one injection point every 5mm on the 3 first cm of the vagina and on the posterior part of the introitus.
  Arms: HA Injection Group

SUMMARY:
Many studies have shown that locoregional treatment (surgery, radiotherapy) and systemic treatment (endocrine therapy and chemotherapy) for breast cancer (BC) may impact sexuality by causing physical and/or psychological damages.

Approximately 50-75 % of BC survivors suffer from vulvovaginal atrophy (VVA). The earliest symptoms of VVA are decreased vaginal lubrication, followed by other vaginal and urinary symptoms, such as burning, itching, bleeding, leucorrhoea, dyspareunia and dysuria symptoms. Various surveys have shown that VVA symptoms lead to female sexual disorder and on their partners through sexual unsatisfactory. However, it appears that sexuality is a little discussed topic during the follow-up of BC survivors. Most of patients relate a poor satisfaction with information and counselling related to sexuality and vaginal health, which are denied by many practitioners.

Patients treated for BC cannot find relief in hormonal replacement therapy (HRT), which is considered the gold standard treatment for VVA symptoms. The usual treatments for these women are topics such as ovula or gel (lubricant, hyaluronic acid (HA)…) with however, a short term effect even when these topics are applied regularly and correctly during at least 2 to 3/weeks.In the literature, there is a significant impact on VVA at one month but later data are lacking . Moreover, patients' compliance and daily application are paramount of importance for efficacy that could disappear when the treatment is stopped.

No randomized controlled trial has compared this treatment to innovative strategies. In this context, it is important to establish management strategies for VVA and sexual disorder after BC.

Our objective is to assess prevalence rate of VVA among breast cancer survivors after the loco regional treatment and chemotherapy, and to compare the efficacy of innovative treatments namely, new biophysical inductor (Laser CO2) and chemical bio inductor (Hyaluronic acid injections) treatments to the efficacy of standard non-hormonal topic treatment for improving the VVA and the quality of sexual life on a long-term.

DETAILED DESCRIPTION:
An open-label multicentre controlled trial randomized in 3 parallel groups (1:1:1) to assess the one-year superiority of bio physical inductor (C02 laser, D0 and M6, group laser) compared to the standard treatment currently recommended (Mucogyne, 2 times a week for one year, control group) in the one hand, and of chemical bio inductor (Desirial, injection of 1 mL of hyaluronic acid in the first 3 cm of the vaginal walls, D0 and M6, HA injection group) compared to the control group in the other hand in BC survivors with VVA, with blinded primary endpoint assessment.

The use of these innovative treatments (lasers and injections) for Vulvovaginal atrophy based on the bio induction and the regenerative medicine could improve the quality of the vaginal mucosa after breast cancer therapy and could be a new strategy for these women who cannot benefit from Hormone Replacement Therapy (HRT). The benefits expected are the improvement of the quality of vulvo-vaginal mucosa and the improvement of the sexual quality of life of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Women who present VVA with a vaginal health index < 15
* 18 years ≤ Age ≤ 75 years
* Patient with non-metastatic breast cancer
* End of loco-regional treatments (surgery+/- radiotherapy) and chemotherapy for 6 months
* Patients with no psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Written consent
* Affiliation to a social security system

Exclusion Criteria:

* Pregnant or breastfeeding woman (A Urinary bHCG will be performed for no menopausal women)
* Vulvo vaginal area showing signs of clinical inflammation and/or viral infection (e.g.: Papilloma, Herpes), bacterial, fungal.
* Abnormal vaginal smear within 3 years before inclusion
* History of vulvo vaginal cancer
* History of Papilloma virus
* History of vaginal herpes
* Use of topical hyaluronic acid application in the month before inclusion
* History of allergy to HA
* Hypersensitivity to the components of Mucogyne®, and Desirial®
* Patients with tendency to develop hypertrophic scars
* No contraception, or no efficient contraception(for women with non-menopausal status)
* Patients under legal protection
* Prisoners
* Participation to another interventional study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 330 (Estimated)
Dates: Start 2021-02-21 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of women free from vulvo-vaginal atrophy on the basis of a vaginal health index (VHI) ≥ 15. | at 12 months

SECONDARY OUTCOMES:
Comparisons among groups of VHI score (absolute and relative changes in the VHI) | Day 0 to 12 months
Female Sexual Distress (FSD) SCALE | Day 0 to 12 months
Evaluation of the pain during treatment (Visual Analogue Scale (EVA)) | Day 0 to 12 months
Rate of adverse effects | Day 0 to 12 months
compliance in the control treatment by the count of forgetfulness during the treatment per topical gel | Day 0 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara HERSANT, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Yazid BELKACEMI, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri-Mondor Hospital, Créteil, France